CLINICAL TRIAL: NCT02713256
Title: An Open Label Study to Evaluate the Safety and Efficacy of 12 Week Treatment With CFZ533 in Patients With Graves' Disease
Brief Title: A Study to Evaluate the Safety and Effect of CFZ533 on Patients With Graves' Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCFZ533X2205; 2015-005564-41 (EudraCT Number)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Graves' Disease
Keywords: Graves' disease; Hyperthyroidism; CFZ533; TSH
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — iscalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CFZ533 10mg/kg (Experimental): CFZ533 intravenously over approximately one hour
  Interventions: Drug: CFZ533

INTERVENTIONS:
Drug: CFZ533 — CFZ533 intravenously over approximately one hour

SUMMARY:
An open label study to evaluate the safety and efficacy of CFZ533 following 12 weeks treatment in patients with Graves' disease

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients 18 to 65 years of age included.
* Women of child-bearing potential must be willing to use highly effective methods of contraception during the study treatment epoch and for 12 weeks after the last study treatment.
* Graves' hyperthyroidism, with the following labs measured at screening:
* TSH<LLN and either FT3>ULN or FT4> ULN and
* TRAb ≥ 2.5 IU/L
* Patients must weigh at least 40 kg to participate in the study

Key Exclusion Criteria:

* History of treatment of Graves' disease with radio-iodine ablation or thyroidectomy and/or current treatment with anti-thyroid drugs (methimazole or propylthiouracil) within one week of starting the study treatment
* History of hyperthyroidism not caused by Graves' disease (e.g. toxic multinodular goiter, autonomous thyroid nodule, or acute inflammatory thyroiditis) and/or history or presence of thyroid storm (fever, profuse sweating, vomiting, diarrhea, delirium, severe weakness, seizures, markedly irregular heartbeat, yellow skin and eyes (jaundice), severe low blood pressure, and coma).
* Previous treatment with a B cell-depleting biologic agent or any other immune-modulatory biologic agent within 5 half-lives (experimental or approved).
* History of recurrent clinically significant infection or of recurrent bacterial infections with encapsulated organisms.
* History of primary or secondary immunodeficiency, including a positive HIV (ELISA and Western blot) test result.
* History or evidence of tuberculosis by either of the following tests:
* Positive PPD skin test (size of induration measured after 48-72 hours, and a positive result is defined as an induration of ≥ 5mm or according to local practice/guidelines) OR
* Positive QuantiFERON TB-Gold test
* Plans for immunization with a live vaccine within a 2-month period before enrollment or during the study period.
* Treatment with immunomodulatory drugs, such as cyclosporine A, methotrexate, and/or cyclophosphamide within 3 months from baseline. Glucocorticosteroid therapy with prednisolone up to 10 mg daily is permitted if patients are on stable dose for more than 3 months before enrollment in the study.
* Pregnant, breastfeeding females, and women of child bearing potential unless they are using highly effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (2):
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Rochester, Minnesota
- Novartis Investigative Site, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Faustino LC, Kahaly GJ, Frommer L, Concepcion E, Stefan-Lifshitz M, Tomer Y. Precision Medicine in Graves' Disease: CD40 Gene Variants Predict Clinical Response to an Anti-CD40 Monoclonal Antibody. Front Endocrinol (Lausanne). 2021 Jun 4;12:691781. doi: 10.3389/fendo.2021.691781. eCollection 2021. PMID 34149627
- [Derived] Kahaly GJ, Stan MN, Frommer L, Gergely P, Colin L, Amer A, Schuhmann I, Espie P, Rush JS, Basson C, He Y. A Novel Anti-CD40 Monoclonal Antibody, Iscalimab, for Control of Graves Hyperthyroidism-A Proof-of-Concept Trial. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz013. doi: 10.1210/clinem/dgz013. PMID 31512728
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=228

RESULTS

PARTICIPANT FLOW:
Groups:
- CFZ533 10 mg/kg: CFZ533 intravenously over approximately one hour
Period: Overall Study
Arm/Group | CFZ533 10 mg/kg
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CFZ533 10 mg/kg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Whose Thyroid Stimulating Hormone (TSH) Levels Normalize After 12 Week Treatment
Description: Normalization of TSH is defined as TSH level greater than 0.35 mU/L after 12 week treatment (Day 85)
Time Frame: 12 week (DAY 85)
Population: Pharmacodynamic (PD) Analysis Set- all patients in the study was included in this analysis set. Patients who discontinue before 4 weeks of treatment for any reason are not counted for the calculation of responders.
Measure: Number; unit: percentage of participants
Arm/Group | CFZ533 10 mg/kg
Number analyzed (Participants) | 13
percentage of participants | 0

2. Primary Outcome: Percentage of Participants Whose Total Triiodothyronine (Total T3) Levels Decrease After 12 Week Treatment
Description: Percentage of participants whose total triiodothyronine (total T3) levels decrease after 12 week treatment. A decrease is when total T3 level is below Upper limit of normal (ULN) ≤ 2.79 nmol/L
Time Frame: 12 week (DAY 85)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CFZ533 10 mg/kg
Number analyzed (Participants) | 13
percentage of participants | 38.5

3. Primary Outcome: Percentage of Participants Whose Free Thyroxine (Free T4) Levels Decrease After 12 Week Treatment
Description: Percentage of participants whose free thyroxine (free T4) levels decrease after 12 weeks of treatment (DAY85). A decrease is when free T4 level is below Upper limit of normal (ULN) ≤ 22.7 pmol/L)
Time Frame: 12 week (DAY 85)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CFZ533 10 mg/kg
Number analyzed (Participants) | 13
percentage of participants | 30.8

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to 36 weeks Day 253.
Arm/Group | CFZ533 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 10 mg/kg (N=15)
TACHYCARDIA (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 10 mg/kg (N=15)
PALPITATIONS (Cardiac disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
DRY MOUTH (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 2
CYSTITIS (Infections and infestations) | 3
SKIN INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
CARDIAC MURMUR (Investigations) | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1
HEADACHE (Nervous system disorders) | 2
INSOMNIA (Psychiatric disorders) | 2
SLEEP DISORDER (Psychiatric disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02713256/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02713256/SAP_001.pdf